CLINICAL TRIAL: NCT03775473
Title: Dosage of Progastrin in Asymptomatic Person Participating in Colon Cancer Screening
Brief Title: PROgastrine COlon DEpistage
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic has made it increasingly difficult for ECS progastrin to ensure clinical research is maintained.
  As a result, the sponsor made the decision to end patient enrollment prematurely.
Sponsor: ECS-Progastrin SA (Industry)
Collaborators: Centre Hospitalier Princesse Grace (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROCODE
Record Dates: First submitted 2018-12-07; First posted 2018-12-14 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Colon Cancer Screening; Healthy Person
Keywords: progastrin; screening; bio-marker; healthy person; early stage

STUDY DESIGN:
Intervention Model Description: Interventional Research, at Risk and Minimal Constraints, Category 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- progastrin (Other): anyone who will participate in colon screening at the Princess Grace Hospital in Monaco and who has signed the informed consent document
  Interventions: Diagnostic Test: progastrin

INTERVENTIONS:
Diagnostic Test: progastrin — PROCODE is an interventional study of category 2 (non-medicinal product), with a minimal risks and restrictions, involving only one blood drawn at the screening of colon cancer.

SUMMARY:
Dosage of progastrin in asymptomatic person participating in colon cancer screening

DETAILED DESCRIPTION:
For anyone who will participate in colon screening at the Princess Grace Hospital of Monaco and who has signed the informed consent document. A blood test will be performed in addition to the screening test to assess the rate of progastrin.

ELIGIBILITY:
Inclusion Criteria:

* participant in colon cancer screening
* signing informed consent

Exclusion Criteria:

* any major medical, psychiatric or addictive illness that would affect the informed consent process
* The consent of a representative is not allowed in this study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
progastrin rate | from 15 days to 2 months (until results are obtained)
  measuring the rate of progastrin in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Georges GARNIER, Principal Investigator — Centre Hospitalier Princesse Grace
Locations (1):
- Centre Hospitalier Princesse Grace, Monaco, Montpellier, MC, France

IPD SHARING:
Plan to Share IPD: No
Monocentric study; No IPD sharing